CLINICAL TRIAL: NCT07321756
Title: Clinical Study on the Application of Presbyopia-correcting Intraocular Lenses in the Surgery of Cataract Patients With Combined Anterior Segment Structural Abnormalities
Brief Title: Evaluating Presbyopia-Correcting IOLs in Complex Cataract Cases With Anterior Segment Abnormalities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-1077
Record Dates: First submitted 2025-12-07; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Lens Diseases
MeSH Terms: conditions — Lens Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unilateral Posterior Chamber Presbyopia-Correcting IOL Implantation Group (Experimental): This arm includes four cohorts of cataract patients with different types of anterior segment structural abnormalities: the lens subluxation group, the chronic anterior uveitis with cataract group, the post-myopic laser corneal surgery with cataract group, and the aphakia with insufficient capsular support group. Patients in each group will undergo unilateral posterior chamber implantation of a suitable type of presbyopia-correcting IOL based on their individual characteristics.
  Interventions: Procedure: Unilateral Posterior Chamber Implantation of Presbyopia-Correcting IOL
- Unilateral Posterior Chamber Monofocal IOL Implantation Group (Active Comparator): This arm includes four cohorts of cataract patients with different types of anterior segment structural abnormalities: the lens subluxation group, the chronic anterior uveitis with cataract group, the post-myopic laser corneal surgery with cataract group, and the aphakia with insufficient capsular support group. Patients in each control group will undergo unilateral posterior chamber implantation of a monofocal IOL of the same brand as that used in the experimental group.
  Interventions: Procedure: Unilateral Posterior Chamber Implantation of Monofocal IOL

INTERVENTIONS:
Procedure: Unilateral Posterior Chamber Implantation of Presbyopia-Correcting IOL — Based on the specific characteristics and needs of each of the four patient groups, a suitable presbyopia-correcting IOL will be selected and precisely implanted unilaterally in the posterior chamber.
  Arms: Unilateral Posterior Chamber Presbyopia-Correcting IOL Implantation Group
Procedure: Unilateral Posterior Chamber Implantation of Monofocal IOL — Each control group will undergo unilateral posterior chamber implantation of the same-brand monofocal IOL as used in the experimental group, following conventional selection criteria.
  Arms: Unilateral Posterior Chamber Monofocal IOL Implantation Group

SUMMARY:
The goal of cataract surgery has evolved from simply restoring sight to providing clear and comfortable full-range vision. Traditionally, monofocal IOLs remain the routine choice for special cases with anterior segment abnormalities-such as lens subluxation, cataract with chronic uveitis, post-laser refractive cataract, and aphakia with insufficient capsular support. However, there is a growing demand among these patients for improved visual quality and spectacle independence.Currently, various presbyopia-correcting IOLs offer distinct advantages, providing more personalized options. The introduction and application of intraoperative optical coherence tomography (iOCT) ensures effective intraoperative monitoring. These advances make the precise implantation of presbyopia-correcting IOLs a promising extension to phacoemulsification in complex cataracts with anterior segment abnormalities.

Nevertheless, their exact benefits regarding visual quality, safety, and patient satisfaction require systematic evaluation through rigorous prospective studies and long-term follow-up. Under strict perioperative management, this study will employ iOCT to monitor the accurate implantation of presbyopia-correcting IOLs and will assess postoperative visual quality and patient satisfaction.

DETAILED DESCRIPTION:
With the evolution of refractive cataract surgery, the goal of treatment has progressed from simple visual rehabilitation to providing clear and comfortable full-range vision through the implantation of functional intraocular lenses (IOLs). Traditionally, monofocal IOLs have been the standard choice for patients with anterior segment abnormalities-such as lens subluxation, cataract with a history of chronic anterior uveitis, post-laser refractive surgery cataract, or aphakia with insufficient capsular support-to minimize adverse optical outcomes. However, these patients, who span a broad age range, increasingly desire high postoperative visual quality and reduced spectacle dependence. Modern presbyopia-correcting IOLs offer advantages in material properties, structural design, and optical performance, improving biocompatibility and reducing visual disturbances such as glare and halos, thereby expanding personalized options. The integration of intraoperative optical coherence tomography (iOCT) further enhances the precision and safety of IOL implantation.

Based on these advancements, the precise implantation of presbyopia-correcting IOLs holds promise for complex cataract cases with anterior segment abnormalities. Nevertheless, their efficacy, safety, and impact on patient satisfaction require systematic evaluation through well-designed prospective studies. This prospective study aims to assess the clinical outcomes of precisely implanted presbyopia-correcting IOLs in patients with complex cataract and anterior segment structural abnormalities, including lens subluxation, chronic anterior uveitis, post-refractive surgery status, and aphakia with inadequate capsular support. Utilizing iOCT for real-time monitoring of anterior segment anatomy, capsular stability, and effective lens position (ELP) during surgery, the study will compare visual quality, safety parameters, and patient satisfaction between presbyopia-correcting IOLs and conventional monofocal IOLs, providing evidence to support individualized IOL selection in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Lens Subluxation Unilateral Implantation Group

   * Patients aged 18-80 years with diagnosed lens subluxation meeting surgical indications for lens surgery, enrolled unilaterally;
   * Informed consent for the study;
   * Ability to comply with full follow-up;
   * Kappa angle <0.5 mm, total higher-order aberration root mean square (HOA RMS) within the central 4-mm corneal zone <1 μm;
   * Mesopic natural pupil diameter between 3.0 mm and 5.5 mm;
   * Expected postoperative astigmatism ≤1.0 D, with target spherical equivalent between 0.00 D and ±0.75 D;
   * Subjective desire to improve full-range visual function.
2. Inactive Long-standing Anterior Uveitis with Cataract Unilateral Implantation Group

   * Patients aged 18-80 years with diagnosed inactive long-standing anterior uveitis (quiet for ≥3 months) and cataract meeting surgical indications for lens surgery, enrolled unilaterally;
   * Centered pupil without significant deformity, with expected postoperative mesopic natural pupil diameter between 2.5 mm and 5.5 mm;
   * Informed consent for the study;
   * Ability to comply with full follow-up;
   * Kappa angle <0.5 mm, total higher-order aberration root mean square (HOA RMS) within the central 4-mm corneal zone <1 μm;
   * Expected postoperative astigmatism ≤1.0 D, with target spherical equivalent between 0.00 D and ±0.75 D;
   * Subjective desire to improve full-range visual function.
3. Post-myopic Laser Corneal Surgery with Cataract Unilateral Implantation Group

   * Patients aged 18-80 years with cataract following prior myopic laser corneal surgery meeting surgical indications for lens surgery, enrolled unilaterally;
   * Informed consent for the study;
   * Ability to comply with full follow-up;
   * Kappa angle <0.5 mm, total higher-order aberration root mean square (HOA RMS) within the central 4-mm corneal zone <1 μm;
   * Mesopic natural pupil diameter between 3.0 mm and 5.5 mm;
   * Expected postoperative astigmatism ≤1.0 D, with target spherical equivalent between 0.00 D and ±0.75 D;
   * Subjective desire to improve full-range visual function.
4. Aphakia with Insufficient Residual Capsular Support Unilateral Implantation Group

   * Patients aged 18-80 years with aphakia and insufficient residual capsular support meeting surgical indications for IOL implantation, enrolled unilaterally;
   * Informed consent for the study;
   * Ability to comply with full follow-up;
   * Kappa angle <0.5 mm, total higher-order aberration root mean square (HOA RMS) within the central 4-mm corneal zone <1 μm;
   * Mesopic natural pupil diameter between 3.0 mm and 5.5 mm;
   * Expected postoperative astigmatism ≤1.0 D, with target spherical equivalent between 0.00 D and ±0.75 D;
   * Subjective desire to improve full-range visual function.

Exclusion Criteria:

1. Lens Subluxation Unilateral Implantation Group

   * Patients with coexisting ocular developmental anomalies such as microphthalmos or microcornea.
   * Patients with severe or progressive ocular diseases (e.g., glaucoma, diabetic retinopathy, macular degeneration) or severe optic nerve disorders.
   * Patients with other organic ocular pathologies, including pathologic high myopia with fundus changes, significant pupillary abnormalities (excessively large or small pupils), severe corneal disease or scarring, high irregular astigmatism, chronic uveitis, or severe amblyopia.
   * Patients with lens disorders other than subluxation and cataract.
   * Patients experiencing intraoperative complications that may affect IOL position and outcome (e.g., posterior capsule rupture, iris prolapse)
   * Patients with a history of prior ocular surgery such as corneal refractive laser surgery, glaucoma surgery, or vitrectomy.
2. Inactive Long-standing Anterior Uveitis with Cataract Unilateral Implantation Group

   * Patients with active systemic autoimmune diseases, or any systemic disease history or medication use known to significantly affect vision.
   * Patients with coexisting ocular developmental anomalies such as microphthalmos or microcornea.
   * Patients with severe or progressive ocular diseases (e.g., glaucoma, diabetic retinopathy, macular degeneration) or severe optic nerve disorders.
   * Patients with other organic ocular pathologies, including pathologic high myopia with fundus changes, severe corneal disease or scarring, high irregular astigmatism, active uveitis, significant abnormalities of the lens capsule or zonules, or severe amblyopia.
   * Patients experiencing intraoperative complications that may affect IOL position and outcome (e.g., posterior capsule rupture, iris prolapse).
   * Patients with a history of prior ocular surgery such as corneal refractive laser surgery, glaucoma surgery, or vitrectomy.
3. Post-myopic Laser Corneal Surgery with Cataract Unilateral Implantation Group

   * Patients with coexisting ocular developmental anomalies such as microphthalmos or microcornea.
   * Patients with severe or progressive ocular diseases (e.g., glaucoma, diabetic retinopathy, macular degeneration) or severe optic nerve disorders.
   * Patients with other organic ocular pathologies, including pathologic high myopia with fundus changes, significant pupillary abnormalities (excessively large or small pupils), severe corneal disease, high irregular astigmatism, chronic uveitis, significant abnormalities of the lens capsule or zonules, or severe amblyopia.
   * Patients experiencing intraoperative complications that may affect IOL position or outcome (e.g., posterior capsule rupture, iris prolapse).
   * Patients with a history of prior ocular surgery such as glaucoma surgery or vitrectomy.
4. Aphakia with Insufficient Residual Capsular Support Unilateral Implantation Group

   * Patients with coexisting ocular developmental anomalies such as microphthalmos or microcornea.
   * Patients with severe or progressive ocular diseases (e.g., glaucoma, diabetic retinopathy, macular degeneration) or severe optic nerve disorders.
   * Patients with other organic ocular pathologies, including pathologic high myopia with fundus changes, significant pupillary abnormalities (excessively large or small pupils), severe corneal disease or scarring, high irregular astigmatism, chronic uveitis, or severe amblyopia.
   * Patients experiencing intraoperative complications that may affect IOL position or outcome (e.g., iris prolapse).
   * Patients with a history of prior ocular surgery such as corneal refractive laser surgery, glaucoma surgery, or posterior vitrectomy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Uncorrected Distance Visual Acuity (UDVA) | Preoperatively, and postoperatively at 1 day, 1 week, 1 month, and 3 months.
  Visual acuity measured at distance（at 5m) without correction.
Effective Lens Position (ELP) | Baseline, and postoperatively at 1 month, and 3 months
  ELP determined by IOLMaster 700, anterior segment optical coherence tomography (AS-OCT), and anterior segment photography.
Contrast sensitivity (at 2.5 m) | Preoperatively, and postoperatively at 1 week, 1 month, and 3 months
  Uncorrected binocular contrast sensitivity was recorded under mesopic, mesopic with glare, photopic, and photopic with glare conditions at spatial frequencies of 3, 6, 12, and 19 cpd.）
Defocus curve (at 5 m) | Preoperatively, and postoperatively at 1 month and 3 months
  Defocus curves were obtained monocularly and binocularly under uncorrected vision with a micro-monovision setup. Acuity was recorded across 13 refractive intervals from +2.00 D to -4.00 D in 0.50 D decrements.
Optical visual quality | Postoperatively at 1 week, 1 month, and 3 months
  Visual symptoms (glare/halos/starburst) assessed via QoV questionnaire
Visual Function Assessment | Postoperatively at 1 week, 1 month, and 3 months
  Visual Function Index-14 Chinese Version (VF-14-CN) Questionnaire
Best Corrected Visual Acuity (BCVA) | Preoperatively, and postoperatively at 1 day, 1 week, 1 month, and 3 months
  Best Corrected Visual Acuity at distance (at 5m)
Uncorrected Intermediate Visual Acuity (UIVA) | Preoperatively, and postoperatively at 1 day, 1 week, 1 month, and 3 months
  Uncorrected visual acuity (UCVA) at intermediate.
Uncorrected Near Visual Acuity (UNVA) | Preoperatively, and postoperatively at 1 day, 1 week, 1 month, and 3 months
  Uncorrected visual acuity (UCVA) at near (at 40 cm).

SECONDARY OUTCOMES:
Intraocular pressure (IOP) | Preoperatively, and postoperatively at 1 day, 1 week, 1 month, and 3 months
  Intraocular pressure (IOP) measured by non-contact tonometer.(mmHg)
Pupil Diameter | Preoperatively, and postoperatively at 1 day, 1 week, 1 month, and 3 months
  Measuring Pupil Diameter
Ocular B-scan ultrasound | Preoperatively, and postoperatively at 1 month and 3 months
Dry Eye Assessment | Preoperatively, and postoperatively at1 week, 1 month, and 3 months
  Dry eye assessment via Tear Film Break-Up Time (TFBUT)
Fundus assessment | Preoperatively, and postoperatively at 1 week, 1 month, and 3 months
  Fundus assessment via fundus photography and macular optical coherence tomography (OCT).
Endothelial cell density | Preoperatively and postoperatively 1 month
  Endothelial cell density（%）
Frequency of using glasses | Postoperatively at 1 week, 1 month, and 3 months
  Frequency ratings for the use of corrective glasses at a distance, medium range, and close range.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Xu, Phd, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No